CLINICAL TRIAL: NCT02178215
Title: Effect of Holly Mangrove Shower Gel Containing Acanthus Ebracteatus Vahl. on Skin Barrier Function in Atopic Dermatitis Patients
Brief Title: Effect of Holly Mangrove Shower Gel in Atopic Dermatitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Si479/2013
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; skin barrier function; transepidermal water loss; skin pH; stratum corneum hydration; sebum; wrinkle
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo shower gel (Placebo Comparator): •Wash forearm by prepared placebo shower gel twice a day
  Interventions: Other: Placebo shower gel
- Holly Mangrove Shower Gel (Active Comparator): •Wash forearm by Holly Mangrove Showver gel twice a day
  Interventions: Other: Holly Mangrove Shower Gel

INTERVENTIONS:
Other: Placebo shower gel — Wash forearm with placebo shower gel for 10 seconds, twice a day, 2 weeks
  Arms: Placebo shower gel
Other: Holly Mangrove Shower Gel — Wash forearm with Holly Mangrove shower gel containing Acanthus ebracteatus Vahl for 10 seconds, twice a day, 2 weeks
  Arms: Holly Mangrove Shower Gel

SUMMARY:
Atopic dermatitis is a chronic intermittent inflammatory skin disease. Currently, there are many cosmeceutical skin products in which their major action affects skin hydration and skin barrier function. In addition, there are some herbal medication remedies used for the treatment of skin diseases based on the knowledge of Thai traditional medicine. Patients with pruritic rash symptoms who attended the Center of Applied Thai Traditional Medicine, Siriraj Hospital, were prescribed the Holly Mangrove Shower Gel to use and on the follow-up appointment showed significant improvement. Nevertheless, the knowledge of using this herbal medication for treating pruritic skin rash so far has been categorized as folk wisdom and not been confirmed by any clinical-trial study on its efficacy and mechanism of action.

Research teams chose Holly Mangrove Shower Gel containing Acanthus ebracteatus Vahl to act as adjunctive for treating atopic dermatitis. Thus, for the purpose of studying the efficacy of Holly Mangrove Shower Gel containing Acanthus ebracteatus Vahl in improving the skin barrier function in atopic dermatitis.

DETAILED DESCRIPTION:
The investigators team research with patients by separate patients into 2 groups and compare among each other. In the first group use placebo, the other group use Holly Mangrove Shower Gel. To compare outcomes, the investigators will measure transepidermal water loss, stratum corneum hydration, skin pH, sebum and wrinkles after using studied gel.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or above
* Diagnosed as atopic dermatitis (Hanafin and Rajka criteria)
* No active dermatitis within 2 weeks

Exclusion Criteria:

* Pregnancy or lactation
* Any other skin diseases on forearms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Improvement of skin barrier function | baseline, 2 week
  •Measurement of bioengineering property of skin using Tewameter (transepidermal water loss), Corneometer (stratum corneum hydration), pH meter (skin pH), sebumeter (sebum), and visioscan (wrinkle)

SECONDARY OUTCOMES:
Reduction of severity of pruritus | baseline, 2 week
  Evaluation of pruritus by using visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Papapit Tuchinda, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital Mahidol Univeristy, Bangkok, Bangkok, Thailand